CLINICAL TRIAL: NCT06618391
Title: Envafolimab and Recombinant Human Endostatin and Recombinant Human Adenovirus Type 5 Intratumor Local Injection Combined With Systemic Therapy in Patients With Advanced NSCLC :a Prospective, Exploratory Phase II Clinical Study Tudy
Brief Title: Local Injection and Systemic Therapy in the Treatment of NSCLC.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, WuHongbo, Henan Cancer Hospital, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERR-NSCLC-01
Record Dates: First submitted 2024-09-08; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Envafolimab; Recombinant human endostatin; Recombinant Human Adenovirus Type 5; Intratumor local injection; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — envafolimab; Endostatins; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Envafolimab (Experimental): Envafolimab 150 mg Q3W (maximum 2 cycles of intratumoral therapy) was injected intratumorally on days 1 and 8, combined with chemotherapy + Recombinant human endostatin Q3W for 4-6 cycles;
  Interventions: Drug: Envafolimab
- Recombinant human endostatin (Experimental): Intratumoral injection of Recombinant human endostatin15mg Q3W (maximum 2 cycles of intratumoral therapy) on Days 1 and 8; combined chemotherapy + Enbrelizumab Q3W for 4-6 cycles.
  Interventions: Drug: Recombinant human endostatin
- Recombinant human adenovirus type 5 (Experimental): 1.0 ml of recombinant human adenovirus type 5 injected intratumorally on days 1 and 8, Q3W (maximum 2 cycles of intratumoral therapy); combined chemotherapy + envolumab, Q3W, 4-6 cycles of treatment.
  Interventions: Drug: recombinant human adenovirus type 5

INTERVENTIONS:
Drug: Envafolimab — Envolimab :150 mg/time, intratumoral injection, at least 5 sites; Recombinant human endostatin： Q3W for 4-6 cycles，Maintenance therapy 210 mg ,CIV 72 hours ,administered as continuous intravenous pump, administered on Day 1 of each cycle; Docetaxel: 60-75 mg/m2, D1, Q3W,for 4-6 cycles，intravenous drip.
  Other Names: PD-L1
  Arms: Envafolimab
Drug: Recombinant human endostatin — Recombinant human endostatin: 15mg/time, intratumoral injection, at least 5 sites; Envolimab :Maintenance therapy 300 mg, Q3W for 4-6 cycles，, subcutaneous injection; administered on Day 1 of each cycle; Docetaxel: 60-75 mg/m2, D1, Q3W,for 4-6 cycles，intravenous drip.
  Other Names: Endostar
  Arms: Recombinant human endostatin
Drug: recombinant human adenovirus type 5 — Recombinant Human Adenovirus Type 5: 1.0ml/time, intratumoral injection, at least 5 sites; Envolimab :Maintenance therapy 300 mg, Q3W for 4-6 cycles，, subcutaneous injection; administered on Day 1 of each cycle; Docetaxel: 60-75 mg/m2, D1, Q3W,for 4-6 cycles，intravenous drip.
  Other Names: OncorineR
  Arms: Recombinant human adenovirus type 5

SUMMARY:
This study is a prospective, exploratory Phase II clinical study aimed at evaluating the safety and efficacy of Envafolimab and recombinant human endostatin and Recombinant Human Adenovirus Type 5 Intratumor local injection combined with systemic therapy in patients with locally advanced or advanced non-small cell lung cancer(NSCLC).

DETAILED DESCRIPTION:
This study is a prospective, exploratory Phase II clinical study aimed at evaluating the safety and efficacy of Envafolimab and recombinant human endostatin and Recombinant Human Adenovirus Type 5 Intratumor local injection combined with systemic therapy in patients with locally advanced or advanced non-small cell lung cancer(NSCLC).

Patients with pathologically confirmed unresectable locally advanced/advanced NSCLC with atelectasis were screened and eligible subjects were randomized to receive local intratumoral injection of envolumab/Endostar/recombinant human adenovirus type 5 H101 combined with systemic therapy after signing informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate and sign the informed consent form；
2. ≥ 18 years old; Both men and women are eligible；
3. Histologically or cytologically confirmed advanced or metastatic locally advanced, advanced (Stage IIIB, IIIC, or IV) NSCLC without mutations in driver gene testing;
4. Patients with recurrent or metastatic NSCLC who have previously failed first-line standard therapy;
5. According to Response Evaluation Criteria in Solid Tumors (RECIST1.1), there should be at least one measurable lesion as a target lesion, and the measurable lesion should not have received local therapy such as radiotherapy;
6. Atelectasis Radiographically assessed atelectasis with at least one lobe;
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
8. Expected survival ≥3 months;
9. Major organ functions within 7 days prior to treatment meeting the following criteria:(1) Blood routine examination criteria (without blood transfusion within 14 days) : ① Hemoglobin (HB) ≥90g/L; ② absolute neutrophil count (ANC) ≥1.5×10^9/L; ③ Platelet (PLT) ≥80×10^9/L. (2) Biochemical examination should meet the following criteria: ① Total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); ② Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5×ULN, if accompanied by liver metastasis, ALT and AST≤5×ULN; ③ Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr)≥60ml/min; ④ Serum albumin ≥35g/L. (3) Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF)≥lower limit of normal (50%).
10. For female subjects of childbearing potential, a negative urine or serum pregnancy test should be obtained 3 days prior to receiving the first dose of study drug;
11. Subject and subject sexual partner need to use contraceptive measures (eg intrauterine device, contraceptive pill , or condom) during the study treatment period and for 6 months after the end of the study treatment period;

Exclusion Criteria:

1. Severe metamorphosis/allergic reaction to humanized antibodies or fusion proteins;
2. Known hypersensitivity to Endostar or any component of the antibody formulation;
3. Diagnosis of immunodeficiency or ongoing systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of study, physiological doses of glucocorticoids (≤ 10 mg/day prednisone or equivalent) are permitted;
4. Exclude subjects with active, known, or suspected autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitaritis, vasculitis, nephritis, hypothyroidism, including but not limited to these diseases or syndromes). Subjects who have type 1 diabetes, hypothyroidism requiring hormone replacement therapy, skin conditions that do not require systemic treatment (e.g., vitiligo, psoriasis, or hair loss), or conditions that are not expected to recur in the absence of external triggers may be enrolled;
5. Patients with severe heart disease, including congestive heart failure, uncontrolled high-risk arrhythmia, unstable angina pectoris, myocardial infarction, severe heart valve disease;
6. Patients who have previously received targeted therapy with vascular endothelial growth inhibitors, such as bevacizumab, Sunitinib, sorafenib, imatinib, Famitinib, Regafenib, Apatinib, androtinib, etc.
7. Systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or mitomycin C within 6 weeks prior to receiving trial drug) planned within 4 weeks prior to group assignment or during this study. Expansion field radiotherapy (EF-RT) within 4 weeks before grouping or limited field radiotherapy to assess tumor lesions within 2 weeks before grouping;
8. Active hepatitis B (HBV DNA ≥ 2000IU/ml or 104copies/ml), hepatitis C (hepatitis C antibody positive and HCV-RNA higher than the lower limit of assay);
9. Active pulmonary tuberculosis (TB) infection was judged based on chest X-ray, sputum examination, and clinical examination. Patients with a history of active pulmonary tuberculosis infection within the previous year, even if treated, were excluded; patients with a history of active pulmonary tuberculosis infection more than 1 year ago, unless the course and type of anti-tuberculosis treatment previously used were proven to be appropriate.
10. Patients with brain metastases accompanied by symptoms or symptom control time less than 2 months;
11. Received significant surgical treatment, open biopsy, or obvious traumatic injury within 28 days prior to grouping;
12. imaging showed that the tumor has invaded important blood vessels or the investigator judged that the tumor is likely to invade important blood vessels during the subsequent study period and cause fatal bleeding;
13. regardless of severity, patients with any signs of bleeding constitution or medical history; within 4 weeks before grouping, patients with any bleeding or bleeding events ≥ CTCAE grade 3, with unhealed wounds, ulcers or fractures;
14. Hyperarterial/venous thrombotic events within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism;
15. According to the investigator 's judgment, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
lung recruitment rate | every 3 weeks during intratumoral treatment in the first two cycles,At the end of Cycle 1and Cycle2 (each cycle is 281days).
  Imaging studies showed that the lesion dissipated or atelectasis was reduced by 50%

SECONDARY OUTCOMES:
ORR（Objective response rate） | Assessed every 6 weeks （within 1 year）or every 9 weeks （1 year later）up to disease progression or death or up to 2 years
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR assessed by the investigator according to RECIST version 1.1
DCR（Disease control rate） | Assessed every 6 weeks （within 1 year）or every 9 weeks （1 year later）up to disease progression or death or up to 2 years
  DCR was defined as the percentage of CR+PR+SD assessed by the investigator according to RECIST version 1.1
PFS（Progression-free survival） | Assessed every 6 weeks （within 1 year）or every 9 weeks （1 year later）up to disease progression or death or up to 2 years
  PFS was defined as the time from first dose to first documented disease progression (PD) or death from any cause, whichever occurred first.
OS（Overall survival） | up to 2 years
  OS was defined as the time from first dose to death for any cause
RFS（Recurrence free survival） | Assessed every 6 weeks （within 1 year）or every 9 weeks （1 year later）up to disease progression or death or up to 2 years
  RFS was defined as the time from CR to disease progression (PD) or death or up to years, from any cause, whichever occurred first.
EORTC QLQ-C30 scale | up to disease progression or 2 years
  The European O-rganization for Reasearch and Treatment of Cancer Quality of Life Questionnare-core 30,There are 30 items in total, of which 29 and 30 items are divided into 7 grades, marked as 1-7 points according to the options, and other items are divided into 4 grades, marked as 1-4 points according to the options.High or low score do not mean a better or worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hongbo Wu, M.D., Principal Investigator — Henan Cancer Hospital

IPD SHARING:
Plan to Share IPD: No